CLINICAL TRIAL: NCT03169153
Title: One-month Clinical Comparison of Silicone Hydrogel Monthly Lenses in High Lipid Depositors
Brief Title: Clinical Comparison of Silicone Hydrogel Monthly Lenses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CLL541-P001
Record Dates: First submitted 2017-05-25; First posted 2017-05-30 (Actual); Results first posted 2019-07-25 (Actual); Last update posted 2019-07-25 (Actual); Status verified 2019-05

CONDITIONS: Refractive Error
Keywords: contact lenses; lipids; deposits
MeSH Terms: conditions — Refractive Errors

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Lotrafilcon B, then senofilcon C (Other): Lotrafilcon B contact lenses worn first, followed by senofilcon C contact lenses, as randomized. Each product worn bilaterally (in both eyes) for a total duration of 30 (+ 3) days under a daily wear modality for the specific study period. The lenses will be removed every night and cared for with the subject's habitual lens care solution.
  Interventions: Device: Lotrafilcon B contact lenses; Device: Senofilcon C contact lenses
- Senofilcon C, then lotrafilcon B (Other): Senofilcon C contact lenses worn first, followed by lotrafilcon B contact lenses, as randomized. Each product worn bilaterally (in both eyes) for a total duration of 30 (+ 3) days under a daily wear modality for the specific study period. The lenses will be removed every night and cared for with the subject's habitual lens care solution.
  Interventions: Device: Lotrafilcon B contact lenses; Device: Senofilcon C contact lenses

INTERVENTIONS:
Device: Lotrafilcon B contact lenses — Silicone hydrogel contact lenses used as per their Conformité Européenne (CE) marking
  Other Names: AIR OPTIX® plus HydraGlyde
Device: Senofilcon C contact lenses — Silicone hydrogel contact lenses used as per their Conformité Européenne (CE) marking
  Other Names: ACUVUE® VITA®

SUMMARY:
The purpose of this study is to compare AIR OPTIX® plus HydraGlyde (AOHG) contact lenses to ACUVUE® VITA® (VITA) contact lenses for total lipid uptake (total of surface and bulk uptake) after 30 days of wear by high lipid depositors.

ELIGIBILITY:
Inclusion Criteria:

* Sign Informed Consent;
* Best corrected visual acuity (BCVA) of at least 0.1 logarithm of the minimum angle of resolution (logMAR) in each eye at Visit 1;
* Manifest cylinder less than or equal to 0.75 diopter (D) in each eye at Visit 1;
* Successful current wearer (during the past 2 months for a minimum of 5 days per week and 8 hours per day) of monthly replacement silicone hydrogel lenses within the power range of lens powers available for the screening and study lenses;
* Screening lenses worn 10 hours exhibiting high lipid uptake.

Exclusion Criteria:

* Habitual lens used in an extended wear modality (routinely sleeping in lenses overnight for 1 night per week or more) during the past 2 months;
* Habitually wearing AIR OPTIX AQUA, AIR OPTIX plus HydraGlyde, ACUVUE OASYS®, or ACUVUE VITA as contact lenses during the past 2 months;
* Any anterior segment infection, inflammation, disease or abnormality that contraindicates contact lens wear (within 7 days of enrollment, or current)
* History of herpetic keratitis, corneal surgery, or irregular cornea;
* Any use of systemic or ocular medications for which contact lens wear could be contraindicated, as determined by the Investigator;
* Abnormal ocular conditions or findings, as specified in the protocol;
* Known pregnancy and lactation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Actual)
Dates: Start 2017-09-22 (Actual); Primary Completion 2018-07-19 (Actual); Study Completion 2018-07-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Manager, Medical Clinical Trial Services, Study Director — Alcon Research
Locations (1):
- Alcon Investigative Site, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from 1 study center located in the United Kingdom.
Pre-assignment Details: Of the 114 enrolled, 29 subjects were exited prior to randomization. An additional 4 subjects discontinued after randomization but prior to exposure. This reporting group includes all randomized and exposed subjects (81).
Groups:
- AOHG Then VITA: Lotrafilcon B contact lenses worn first, followed by senofilcon C contact lenses, as randomized. Each product worn bilaterally (in both eyes) for a total duration of 30 (+ 3) days under a daily wear modality for the specific study period. The lenses were removed every night and cared for with the subject's habitual lens care solution.
- VITA Then AOHG: Senofilcon C contact lenses worn first, followed by lotrafilcon B contact lenses, as randomized. Each product worn bilaterally for a total duration of 30 (+ 3) days under a daily wear modality for the specific study period. The lenses were removed every night and cared for with the subject's habitual lens care solution.
Period: Period 1, First 30 Days of Wear
Arm/Group | AOHG Then VITA | VITA Then AOHG
Started (Randomized and exposed) | 42 | 39
Completed | 39 | 35
Not Completed | 3 | 4
Not completed — Lost to Follow-up | 1 | 1
Not completed — Withdrawal by Subject | 2 | 3
Period: Period 2, Second 30 Days of Wear
Arm/Group | AOHG Then VITA | VITA Then AOHG
Started | 39 | 34 (One subject discontinued after completing Period 1 and was not exposed in Period 2.)
Completed | 37 | 32
Not Completed | 2 | 2
Not completed — Adverse Event | 1 | 2
Not completed — Could not attend visit | 1 | 0

BASELINE CHARACTERISTICS:
Population: This analysis population includes all randomized subjects who were exposed to AOHG or VITA lenses (Full Analysis Set).
Groups:
- Overall: Lotrafilcon B and senofilcon C contact lenses worn during Period 1 and Period 2 in a crossover assignment.
Arm/Group | Overall
Number analyzed (Participants) | 81
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.3 (9.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 60
  Male | 21
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Mean Ex-vivo Total Lipid Uptake (Total of Surface and Bulk Uptake) Per Lens
Description: Contact lens was removed aseptically from the eye. Total lipid (fatty deposits) uptake, defined as total amount of lipids (surface and bulk) absorbed/adsorbed and extracted, was measured in micrograms. A lower value indicates better results. Only one lens from each subject contributed to the analysis.
Time Frame: Day 30 after 10 hours of wear, each product
Population: Full Analysis Set with non-missing response
Measure: Mean (Standard Deviation); unit: micrograms (μg)
Groups:
- AOHG: Lotrafilcon B contact lenses worn bilaterally for 30 (+ 3) days under a daily wear modality. The lenses were removed every night and cared for with the subject's habitual lens care solution.
- VITA: Senofilcon C contact lenses worn bilaterally for 30 (+ 3) days under a daily wear modality. The lenses were removed every night and cared for with the subject's habitual lens care solution.
Arm/Group | AOHG | VITA
Number analyzed (Participants) | 59 | 56
micrograms (μg) | 78.1398 (70.7923) | 307.6800 (303.9299)
Statistical Analysis 1: Comparison: AOHG vs VITA; Test type: Superiority; p < 0.0001, Mixed effects repeated measures

ADVERSE EVENTS:
Time Frame: Dispense through study completion, an average of 2.5 months
Description: An adverse event (AE) was defined as any untoward medical occurrence, unintended disease or injury, or untoward clinical signs in subjects, users, or other persons, whether or not related to the study lenses. AEs were obtained through solicited and spontaneous comments from subjects and through observations by the Investigator as outlined in the study protocol.
Groups:
- AOHG: All subjects exposed to lotrafilcon B contact lenses
- VITA: All subjects exposed to senofilcon C contact lenses
Arm/Group | AOHG | VITA
All-Cause Mortality (participants affected / at risk) | 0/76 | 0/78
Serious Adverse Events (participants affected / at risk) | 0/76 | 0/78
Other Adverse Events (participants affected / at risk) | 0/76 | 0/78

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right of prior review of any publication or presentation of information related to the study.

DOCUMENTS (2):
  • Study Protocol (2017-12-07): https://cdn.clinicaltrials.gov/large-docs/53/NCT03169153/Prot_000.pdf
  • Statistical Analysis Plan (2018-07-03): https://cdn.clinicaltrials.gov/large-docs/53/NCT03169153/SAP_001.pdf